CLINICAL TRIAL: NCT02891265
Title: Smoking Cessation Intervention Within the Fracture Clinic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study stopped due to the difficulty in patient compliance for follow up visits
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20130239-01H
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Focus: Smoking Cessation as it Relates to Fracture Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (No Intervention): Group A - smoking cessation with no assistance
- Group B (Placebo Comparator): Group B - smoking cessation with the addition of a smoking cessation patch
  Interventions: Behavioral: Smoking cessation patch

INTERVENTIONS:
Behavioral: Smoking cessation patch — To compare the smoking cessation outcome in patients with fractures with or without the help of smoking cessation patches.
  Arms: Group B

SUMMARY:
Tobacco use is the leading preventable cause of death contributing to more than 5 million estimated deaths per year globally. The longterm negative effects of smoking are well established. Complications due to smoking, from an orthopaedic perspective include impair bone and wound healing, and increased risk of infection and osteomyelitis.

The primary outcome of this research is smoking cessation in patients attending the orthopaedic fracture clinic. This is a unique environment whereby previously healthy patients are faced with the impact of disability. This impetus to abstain from the benefit of fracture outcomes provides an opportunity for previously unattained early intervention and thus a greater potential for decreased patient morbidity and mortality. Furthermore it is a high volume clinic that, given the unique nature of traumatic injuries consists of a high proportion of males, ages 24-34 years old, obliged to follow up. This population is traditionally regarded as unattainable from primary prevention smoking cessation strategies. The investigators hypothesize that The Ottawa Hospital Fracture Clinic will serve as an effective environment to employ established primary prevention smoking cessation interventions, reducing the incidence of complications associated with fracture and surgical healing, and result in greater long-term cessation rates.

DETAILED DESCRIPTION:
Tobacco use is the leading preventable death contributing to more than 5 million estimated deaths per year globally.1 Nicotine is a highly addictive substance and tobacco remains the only legal product that, when used as intended, kills. The long term negative effects of smoking are well established.

Ten percent of all current and former smokers live with chronic disease. Among current smokers who are ill, the most prevalent conditions are chronic bronchitis, emphysema, and myocardial infarction.2 Moreover complications due to smoking from an orthopaedic perspective are well established. With respect to orthopaedic trauma literature, smoking impairs osteoblastic function, and propagates vasoconstriction resulting in delayed or non -unions.3 Its use has a 3-6 fold increased risk of intra- operative pulmonary complications, impairs wound healing4, healing of bone, soft tissues, and can lead to flap necrosis. 4-7 Furthermore smokers are twice as likely to develop an infection and 3.7 times as likely to develop osteomyelitis8.

Smoking cessation programs are essential in achieving a sustainable health care system. Health care costs for smokers at a given age are as much as 40 percent higher than those for non smokers. 9 The cost of treatment of tobacco related illness in British Columbia in 2004 was estimated to be 500 million CDN dollars. The total annual cost of treatment for conditions related to second hand smoke exposure in North Carolina and Minnesota in 2006 alone were estimated to be greater than 290 and 225 million US dollars respectively. 10, 11

The role of the healthcare practitioner has been recognized as of paramount importance in smoking cessation. These programs rely on the Transtheoretical Model of patient behavioral change. In order to maximize intervention a clinician is to provide counseling, motivation, education, monitoring, and empathy to personalized smoking cessation intervention programs with extended assistance and follow-up12. Multiple fields of medicine have established smoking cessation programs either pre-operatively or during hospitalization. Randomized control trials (RCTs) of hospitalized cardiac patients have exhibited decreased rates of non fatal infarctions, and re-operation, reduced risk and rates of mortality.13 A systematic review revealed 8 pre- operative RCTs that have been performed to date across multiple surgical disciplines with a total of 1156 enrolled patients. Their strategies for counseling and follow up varied. All had more than 20% loss to follow up and this was limited to a maximum of 12 months. However there was a significant decrease in post-operative complications and cessation was maintained at the 12 month follow up.14

Despite the availability of smoking cessation interventions, traditionally they have been underutilized, in part due to frustration, lack of clinician training and organizational support, especially in Orthopaedic Surgery12. Only a single randomized control trial within the setting of an acute fracture clinic has been published to date.15 This multicentred trial in Sweden utilized a standardized 6 week cessation program with nicotine replacement therapy if the patient in the intervention group desired. It captured only 18% of the potential candidates and was limited to a 12 week follow up. Long term cessation rates were not evaluated.

The acute fracture clinic is a unique environment to establish a smoking cessation program in order to achieve primary prevention. Previously healthy patients are faced with the impact of disability and a unique relationship based on trust is established between patients and their surgeons. Given the negative orthopaedic outcomes associated with smoking aforementioned, patients present as an engaged audience, faced with the possibility of chronic disability (poor surgical/fracture outcome) attributed to the continuation of smoking habits. This impetus to abstain for the benefit of fracture outcomes provides a window of opportunity for previously unattained early intervention and thus a greater potential for decreased patient morbidity and mortality. Furthermore, the acute fracture clinic is a high volume clinic whereby as many as 100 patients may visit per clinic per day (patients from regions within the Champlain Local Health Integration Network [LHIN] where smoking prevalence is as high as 30%). Given the unique nature of traumatic injuries, this population consists of a high proportion of males, ages 24-34 years old, who are obliged to follow up for fracture care. This population (24-35 year old males) is traditionally regarded as unattainable for primary prevention smoking cessation strategies.

Primary prevention strategies are paramount from a public health perspective. In targeting a well established smoking cessation campaign in a fracture clinic with the partnership from the University of Ottawa Heart Institute's Division of Prevention and Rehabilitation, patients will be provided expert cessation strategies before the onset of smoking relating disease. The benefits of which extend beyond the patient to their families. The ultimate goal of this project is to develop an intervention model that can be cost effective and universally applied to all orthopaedic clinics within North America. A great potential exists to increase smoking cessation rates, and decrease orthopaedic trauma smoking related morbidity, long term smoking related morbidity, mortality and health care costs.

ELIGIBILITY:
Inclusion Criteria:

patients greater than 18 years patients sustained an injury resulting in a fracture date of recruitment is the initial clinic/consultation/post operative visit. clinic visit is within and including 14 days from initial date of injury or operation

Exclusion Criteria:

Patients presenting to the fracture clinic that:

* Do not meet inclusion criteria
* Are currently following cessation therapy
* Cannot understand or read English or French
* Have abused alcohol within the last six months
* Have abused illicit drugs within the last six months
* Are Pregnant or breast feeding
* Have sustained a pathologic fracture

Definitions

Fractures:

Following fractures are considered one fracture

* Single or combination of fractures involving hand including and distal to proximal row carpal bones
* Single or combination of fractures involving foot including and distal to the midfoot
* Fractures involving radius and ulna presenting at the same level (ie. Distal,diaphyseal, or proximal as per AO classification)
* Fractures involving tibia and fibula presenting at the same level (ie. Distal,diaphyseal, or proximal as per AO classification)

Polytrauma:

Defined as traumatic incident that has resulted in injury to more than just the MSK system at time of index injury

Spinal Trauma:

Defined as sustaining fracture, subluxation, dislocation, disc herniation or neurologic deficit attributed o spinal injury at time of index injury

Neurovascular Compromise:

Defined as complete loss of motor or cutaneous sensation loss at time of index injury

Illicit substance/drug abuse:

Defined as use of illicit substance or non prescribed narcotic within six months of injury

Alcohol Abuse:

Defined as use of alcohol and positive CAGE questionnaire screening

Pathologic/Insufficiency Fracture:

Fracture secondary to osteoporosis/osteopenia, malignant or non malignant lesion, bisphosphonate use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-04; Primary Completion 2021-01 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Comparison of Rates between no intervention and intervention | 5 yr total
  Spontaneous smoking cessation rates within the orthopaedic trauma population (first cohort) are presently unknown within the literature, however hypothesized to be low. The investigators anticipate a greater than 30% long term cessation rate upon implementation of this model, as compared to its previous implementation in different patient settings. A significant decrease in orthopaedic trauma complications, and long term decreased smoking related morbidity and mortality is expected. The primary outcome of this study will be a comparison of long-term smoking cessation rates between the two cohorts of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Werier, Dr., Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - The Ottawa Hospital- Civic campus, Ottawa, Ontario